CLINICAL TRIAL: NCT00482339
Title: PCR-Based Detection of Bacterial Agents in Platelet Concentrates and Whole Blood (First Study)
Brief Title: PCR-Based Detection of Bacterial Agents in Platelet Concentrates and Whole Blood
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Jena (Other)
Other Study IDs: ITM-Jena-935035-1
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Last update posted 2007-06-05 (Estimated); Status verified 2007-05

CONDITIONS: Healthy
Keywords: bacterial contamination; platelet concentrates; blood donation; looxster; pureprove; bacterial genomic DNA; bacterial contamination of platelet concentrates; Preparation of "bacterial DNA" in blood; comparison of blood culture versus NAT

STUDY DESIGN:
Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Using methods of molecular biology bacteria can be detected in blood. In comparison to conventional blood cultures "bacterial DNA" is isolated using a new sample preparation system in platelet apheresis concentrates and in the predonation whole blood of donors.

DETAILED DESCRIPTION:
Bacterial contamination of platelet concentrates is discussed worldwide and according to literature occuring in 1:1000 to 1:5000 concentrates. Bacterial contaminated concentrates can in fact cause severe infections in patients. therefore this study initially intends to detect contamination with "bacterial DNA" in platelet aphereses concentrates. All sample donations are also examined by blood culture for contamination. To exclude already existing "infection" of the donor one tube of whole blood is taken in addition to the other legally required samples for the production of pharmaceutical medicine. All samples are anonymised before passed on for analysing.

ELIGIBILITY:
Inclusion Criteria:

* healthy platelet apheresis donor

Exclusion Criteria:

* Missing health clearance for blood donation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2007-06; Study Completion 2009-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Dagmar Barz, Prof Dr med., Study Director — University Hospital Jena, Germany
Locations (1):
- Institute for Transfusion Medicine, University Hospital Jena, Jena, Thuringia, Germany